CLINICAL TRIAL: NCT02185534
Title: An Open-label, Randomised, Three-way Crossover Study in Healthy Subjects to Assess the Bioequivalence of European Source Generic Clopidogrel Tablets and US and Japanese Source Branded Clopidogrel (Plavix®) Tablets.
Brief Title: Clopidogrel Bioequivalence Study in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: D5130C00131
Record Dates: First submitted 2014-07-04; First posted 2014-07-09 (Estimated); Results first posted 2015-11-30 (Estimated); Last update posted 2016-06-22 (Estimated); Status verified 2016-05

CONDITIONS: Bioequivalence, AUC, Cmax, Pharmacokinetics
Keywords: Clopidogrel, Zyllt, Plavix, Phase I, Healthy Subjects, Pharmacokinetics, Bioequivalence
MeSH Terms: interventions — Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- European clopidogrel tablets, 75 mg (Experimental): Treatment A: a single oral dose of clopidogrel 75 mg film-coated tablet (Zyllt, KRKA - test)
  Interventions: Drug: Clopidogrel
- Japanese clopidogrel tablets, 75 mg (Active Comparator): Treatment B: a single oral dose of clopidogrel 75 mg film-coated tablet (Plavix®, Brystol-Myer Squibb,Sanofi-Aventis, reference)
  Interventions: Drug: Clopidogrel
- US clopidogrel tablets, 75 mg (Active Comparator): Treatment C: a single oral dose of clopidogrel 75 mg film-coated tablet (Plavix®, Sanofi-Aventis, reference)
  Interventions: Drug: Clopidogrel

INTERVENTIONS:
Drug: Clopidogrel — European clopidogrel tablets, 75 mg (test) versus Japanese clopidogrel tablets, 75 mg (reference); European clopidogrel tablets, 75 mg (test) versus US clopidogrel tablets, 75 mg (reference)
  Other Names: Zyllt; Plavix

SUMMARY:
This study will be an open-label, randomised, three-way crossover study in healthy male and female subjects, performed at a single centre. The objective of the study is to assess the bioequivalence between one test formulation (Clopidogrel 75 mg tablet (commercial blister from KRKA) and two reference formulations (Clopidogrel 75 mg tablet [Plavix, sourced in US and Japan]).

DETAILED DESCRIPTION:
Study to evaluate the bioequivalence of orally administered European source clopidogrel tablets and US and Japanese source clopidogrel tablets.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects aged 18 to 55 years with suitable veins for cannulation or repeated venepuncture.
* Females must have a negative pregnancy test at screening and on each admission to the clinical unit, must not be lactating and

  • if of non child-bearing potential, confirmed at screening by fulfilling one of the following criteria:
* Post-menopausal defined as amenorrhoea for at least 12 months or more following cessation of all exogenous hormonal treatments and follicle-stimulating hormone (FSH) levels in the post-menopausal range.
* Documentation of irreversible surgical sterilisation by hysterectomy, bilateral oophorectomy or bilateral salpingectomy but not tubal ligation.

  • if of child-bearing potential and are sexually active must use, with their partner, 2 approved methods of highly effective contraception from the time of IMP administration until 3 months after the last dose of IMP.
* Have a body mass index between 18,5 and 29.9 kg/m2 inclusive and weigh at least 50 kg and no more than 100 kg inclusive.
* Be able to understand, read and speak the German language.

Exclusion criteria

* History of any clinically significant disease or disorder which, in the opinion of the Investigator, may either put the potential subject at risk because of participation in the study, or influence the results or the potential subject's ability to participate in the study.
* Current smokers or those who have smoked or used nicotine products within the previous 3 months.
* History of haemophilia, von Willebrand's disease, lupus anticoagulant, or other diseases/syndromes that can either alter or increase the propensity for bleeding.
* A personal history of vascular abnormalities including aneurysms; a personal history of severe haemorrhage, haematemesis, melena, haemoptysis, severe epistaxis, severe thrombocytopenia, intracranial haemorrhage; or rectal bleeding within 1 year prior to screening; or history suggestive of peptic ulcer disease; or at the discretion of the Investigator.
* Use of aspirin, ibuprofen, NSAIDS, or any other drug known to increase the propensity for bleeding for 2 weeks before randomisation.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 144 (Actual)
Dates: Start 2014-08; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rainard Fuhr, Dr. med., Principal Investigator — PAREXEL International GmbH, Berlin; Glenn Carlson, MD, Study Director — AstraZeneca, Wilmington, US
Locations (1):
- Research Site, Berlin, Germany

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants recruited at PAREXEL Early Phase Clinical Unit Berlin, Germany between August 2014 and September 2014.
Pre-assignment Details: 84 participants recruited; 144 screened, 60 excluded (59 did not meet inclusion criteria and 1 refused participation)
Groups:
- First European, Then Japanese, Then US Clopidogrel: A single oral dose of clopidogrel 75 mg filmcoated tablet (Zyllt, KRKA
  - test) in Period 1; a single oral dose of clopidogrel 75 mg filmcoated tablet (Plavix®, Brystol-Myer Squibb, Sanofi- Aventis, reference) in Period 2; a single oral dose of clopidogrel 75 mg filmcoated tablet (Plavix®, Sanofi- Aventis, reference) in Period 3
- First European, Then US, Then Japanese Clopidogrel: A single oral dose of clopidogrel 75 mg filmcoated tablet (Zyllt, KRKA - test) in Period 1; a single oral dose of clopidogrel 75 mg filmcoated tablet (Plavix®, Sanofi-Aventis, reference) in Period 2; a single oral dose of clopidogrel 75 mg filmcoated tablet (Plavix®, Brystol-Myer Squibb, Sanofi- Aventis, reference) in Period 3
- First Japanese, Then European, Then US Clopidogrel: A single oral dose of clopidogrel 75 mg filmcoated tablet (Plavix®, Brystol-Myer Squibb, Sanofi-Aventis, reference) in Period 1; a single oral dose of clopidogrel 75 mg filmcoated tablet (Zyllt, KRKA - test) in Period 2; a single oral dose of clopidogrel 75 mg filmcoated tablet (Plavix®, Sanofi- Aventis, reference) in Period 3
- First Japanese, Then US, Then European Clopidogrel: A single oral dose of clopidogrel 75 mg filmcoated tablet (Plavix®, Brystol-Myer Squibb, Sanofi- Aventis, reference) in Period 1; a single oral dose of clopidogrel 75 mg filmcoated tablet (Plavix®, Sanofi-Aventis, reference) in Period 2; a single oral dose of clopidogrel 75 mg filmcoated tablet (Zyllt, KRKA - test) in Period 3
- First US, Then European, Then Japanese Clopidogrel: A single oral dose of clopidogrel 75 mg filmcoated tablet (Plavix®, Sanofi- Aventis, reference) in Period 1, a single oral dose of clopidogrel 75 mg filmcoated tablet (Zyllt, KRKA - test) in Period 2; a single oral dose of clopidogrel 75 mg filmcoated tablet (Plavix®, Brystol-Myer Squibb, Sanofi- Aventis, reference) in Period 3
- First US, Then Japanese, Then European Clopidogrel: A single oral dose of clopidogrel 75 mg filmcoated tablet (Plavix®, Sanofi- Aventis, reference) in Period 1; a single oral dose of clopidogrel 75 mg filmcoated tablet (Plavix®, Brystol-Myer Squibb, Sanofi- Aventis, reference) in Period 2; a single oral dose of clopidogrel 75 mg filmcoated tablet (Zyllt, KRKA - test) in Period 3
Period: First Period
Arm/Group | First European, Then Japanese, Then US Clopidogrel | First European, Then US, Then Japanese Clopidogrel | First Japanese, Then European, Then US Clopidogrel | First Japanese, Then US, Then European Clopidogrel | First US, Then European, Then Japanese Clopidogrel | First US, Then Japanese, Then European Clopidogrel
Started | 14 | 14 | 14 | 14 | 14 | 14
Completed | 14 | 14 | 14 | 13 | 14 | 14
Not Completed | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 0
Period: First Washout Period
Arm/Group | First European, Then Japanese, Then US Clopidogrel | First European, Then US, Then Japanese Clopidogrel | First Japanese, Then European, Then US Clopidogrel | First Japanese, Then US, Then European Clopidogrel | First US, Then European, Then Japanese Clopidogrel | First US, Then Japanese, Then European Clopidogrel
Started | 14 | 14 | 14 | 13 | 14 | 14
Completed | 13 | 14 | 14 | 13 | 13 | 13
Not Completed | 1 | 0 | 0 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 1
Period: Second Period
Arm/Group | First European, Then Japanese, Then US Clopidogrel | First European, Then US, Then Japanese Clopidogrel | First Japanese, Then European, Then US Clopidogrel | First Japanese, Then US, Then European Clopidogrel | First US, Then European, Then Japanese Clopidogrel | First US, Then Japanese, Then European Clopidogrel
Started | 13 | 14 | 14 | 13 | 13 | 13
Completed | 13 | 14 | 14 | 13 | 13 | 13
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Second Washout Period
Arm/Group | First European, Then Japanese, Then US Clopidogrel | First European, Then US, Then Japanese Clopidogrel | First Japanese, Then European, Then US Clopidogrel | First Japanese, Then US, Then European Clopidogrel | First US, Then European, Then Japanese Clopidogrel | First US, Then Japanese, Then European Clopidogrel
Started | 13 | 14 | 14 | 13 | 13 | 13
Completed | 13 | 14 | 14 | 13 | 13 | 13
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Third Period
Arm/Group | First European, Then Japanese, Then US Clopidogrel | First European, Then US, Then Japanese Clopidogrel | First Japanese, Then European, Then US Clopidogrel | First Japanese, Then US, Then European Clopidogrel | First US, Then European, Then Japanese Clopidogrel | First US, Then Japanese, Then European Clopidogrel
Started | 13 | 14 | 14 | 13 | 13 | 13
Completed | 13 | 14 | 14 | 13 | 13 | 13
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The overall number of baseline participants is 84, as it comprised all randomized subjects, although one subject withdrew consent prior to the first dose. Thus the safety population includes 83 subjects only.
Groups:
- Total: Total of all reporting groups
Arm/Group | First European, Then Japanese, Then US Clopidogrel | First European, Then US, Then Japanese Clopidogrel | First Japanese, Then European, Then US Clopidogrel | First Japanese, Then US, Then European Clopidogrel | First US, Then European, Then Japanese Clopidogrel | First US, Then Japanese, Then European Clopidogrel | Total
Number analyzed (Participants) | 14 | 14 | 14 | 14 | 14 | 14 | 84
Age, Continuous [Mean (Standard Deviation); unit: years] | 33 (9) | 37 (11) | 36 (10) | 35 (8) | 34 (9) | 36 (11) | 35 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 8 | 7 | 4 | 4 | 37
  Male | 7 | 7 | 6 | 7 | 10 | 10 | 47
Race/Ethnicity, Customized [Number; unit: participants]
  Black or African American | 1 | 0 | 0 | 0 | 0 | 0 | 1
  White | 13 | 14 | 13 | 14 | 12 | 13 | 79
  Other | 0 | 0 | 1 | 0 | 2 | 1 | 4
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 2 | 1 | 3
  Not Hispanic or Latino | 14 | 14 | 14 | 14 | 12 | 13 | 81
BMI (Body Mass Index) [Mean (Standard Deviation); unit: kg/m^2] | 23.7 (3.1) | 24.7 (3.5) | 23.4 (2.9) | 24.1 (2.7) | 23.0 (3.1) | 23.9 (3.1) | 23.8 (3.0)

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics of Clopidogrel by Assessment of Area Under the Curve From Time Zero Extrapolated to Infinity (AUC(0-inf))
Description: Comparison of the pharmacokinetic profile in terms of plasma concentration-time curve from time zero extrapolated to infinity, AUC(0-inf), of clopidogrel sourced in Europe and Japan.
Time Frame: 0 hours (pre-dose), as well as at 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24 and 36 hours post-dose
Population: The pharmacokinetic population consisted of 79 subjects, i.e. all subjects in the safety population for whom AUC(0-last) and Cmax could be calculated for clopidogrel for the test treatment (European) and at least one of the reference treatments (Japanese, US). AUC(0-inf) could not be reliably calculated for many of these subjects.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Groups:
- European Clopidogrel Tablets, 75 mg: Treatment A: a single oral dose of clopidogrel 75 mg film-coated tablet Eu(Zyllt, KRKA - test)
- Japanese Clopidogrel Tablets, 75 mg: Treatment B: a single oral dose of clopidogrel 75 mg film-coated tablet (Plavix®, Brystol-Myer Squibb,Sanofi- Aventis, reference)
Arm/Group | European Clopidogrel Tablets, 75 mg | Japanese Clopidogrel Tablets, 75 mg | US Clopidogrel Tablets, 75 mg
Number analyzed (Participants) | 41 | 45 | 38
ng*h/mL | 1.05 (139.0) | 0.992 (117.9) | 1.09 (106.9)
Statistical Analysis 1: Comparison: European Clopidogrel Tablets, 75 mg vs Japanese Clopidogrel Tablets, 75 mg; Test type: Non-Inferiority or Equivalence — The analysis was conducted using an analysis of variance (ANOVA) including fixed effects for treatment, sequence, period and subject within sequence. All pharmacokinetic parameters were log-transformed prior to analysis. Bioequivalence was concluded, when the 90% confidence interval (CI) for the geometric LS mean ratios were fully contained within the predefined equivalence limits of 0.80 to 1.25; Geometric mean ratio = 104.43, 90% CI 2-sided [92.27 to 118.19] — Geometric mean ratio is calculated as A/B, where A= European clopidogrel and B=Japanese clopidogrel
Statistical Analysis 2: Comparison: European Clopidogrel Tablets, 75 mg vs US Clopidogrel Tablets, 75 mg; The analysis was conducted using an analysis of variance (ANOVA) including fixed effects for treatment, sequence, period and subject within sequence. All pharmacokinetic parameters were log-transformed prior to analysis. Bioequivalence was concluded, when the 90% confidence interval (CI) for the geometric LS mean ratios were fully contained within the predefined equivalence limits of 0.80 to 1.25; Test type: Non-Inferiority or Equivalence — Geometric mean ratio is calculated as A/C, where A= European clopidogrel and C=US clopidogrel; Geometric mean ratio = 97.19, 90% CI 2-sided [81.12 to 116.45] — Geometric mean ratio is calculated as A/C, where A= European clopidogrel and C=US clopidogrel

2. Primary Outcome: Pharmacokinetics of Clopidogrel by Assessment of Observed Maximum Plasma Concentration (Cmax)
Description: Comparison of the pharmacokinetic profile in terms of observed maximum plasma concentration, taken directly from the individual concentration-time curve, Cmax, of clopidogrel sourced in Europe and the US.
Time Frame: 0 hours (pre-dose), as well as at 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24 and 36 hours post-dose
Population: The pharmacokinetic population consisted of 79 subjects, i.e. all subjects in the safety population for whom AUC(0-last) and Cmax could be calculated for clopidogrel for the test treatment (European) and at least one of the reference treatments (Japanese, US)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | European Clopidogrel Tablets, 75 mg | Japanese Clopidogrel Tablets, 75 mg | US Clopidogrel Tablets, 75 mg
Number analyzed (Participants) | 79 | 79 | 79
ng/mL | 0.551 (122.6) | 0.511 (150.6) | 0.521 (122.4)
Statistical Analysis 1: Comparison: European Clopidogrel Tablets, 75 mg vs Japanese Clopidogrel Tablets, 75 mg; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Geometric mean ratio = 108.06, 90% CI 2-sided [95.46 to 122.33] — Geometric mean ratio is calculated as A/B, where A= European clopidogrel and B=Japanese clopidogrel
Statistical Analysis 2: Comparison: European Clopidogrel Tablets, 75 mg vs US Clopidogrel Tablets, 75 mg; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Geometric mean ratio = 105.79, 90% CI 2-sided [95.22 to 117.53] — Geometric mean ratio is calculated as A/C, where A= European clopidogrel and C=US clopidogrel

3. Secondary Outcome: Pharmacokinetics of Clopidogrel by Assessment of Area Under the Curve From Time Zero to the Time of Last Quantifiable Concentration (AUC(0-last))
Description: Comparison of the pharmacokinetic profile in terms of the area under the plasma concentration-curve from time zero to the time of last quantifiable clopidogrel or SR26334 concentration, AUC(0-last), of clopidogrel sourced in Europe and the US.
Time Frame: 0 hours (pre-dose), as well as at 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24 and 36 hours post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | European Clopidogrel Tablets, 75 mg | Japanese Clopidogrel Tablets, 75 mg | US Clopidogrel Tablets, 75 mg
Number analyzed (Participants) | 79 | 79 | 79
h*ng/mL | 0.705 (114.8) | 0.751 (116.5) | 0.767 (107.1)
Statistical Analysis 1: Comparison: European Clopidogrel Tablets, 75 mg vs Japanese Clopidogrel Tablets, 75 mg; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Geometric mean ratio = 93.94, 90% CI 2-sided [87.12 to 101.29] — Geometric mean ratio is calculated as A/B, where A= European clopidogrel and B=Japanese clopidogrel
Statistical Analysis 2: Comparison: European Clopidogrel Tablets, 75 mg vs US Clopidogrel Tablets, 75 mg; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Geometric mean ratio = 92.03, 90% CI 2-sided [84.91 to 99.75] — Geometric mean ratio is calculated as A/C, where A= European clopidogrel and C=US clopidogrel

ADVERSE EVENTS:
Time Frame: From screening until follow-up, i.e. up to 7 weeks after the first dose.
Description: Adverse events (AEs) were assigned to the treatment after which they occurred:
  Treatment A: AEs starting at the time of /after dosing of European clopidogrel tablets Treatment B: AEs starting at the time of / after dosing of Japanese clopidogrel tablets Treatment C: AEs starting at the time of / after dosing of US clopidogrel tablets
Groups:
- Total Number of Participants: total number of subjects exposed to any treatment
Arm/Group | European Clopidogrel Tablets, 75 mg | Japanese Clopidogrel Tablets, 75 mg | US Clopidogrel Tablets, 75 mg | Total Number of Participants
Serious Adverse Events (participants affected / at risk) | 0/81 | 0/80 | 0/82 | 0/83
Other Adverse Events (participants affected / at risk) | 19/81 | 18/80 | 22/82 | 38/83
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | European Clopidogrel Tablets, 75 mg (N=81) | Japanese Clopidogrel Tablets, 75 mg (N=80) | US Clopidogrel Tablets, 75 mg (N=82) | Total Number of Participants (N=83)
Headache (Nervous system disorders) | 16 (19) | 15 (17) | 16 (20) | 29 (56)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 3 (3) | 4 (4)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1/2 (2) | 2/2 (2) | 3/4 (4)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Catheter Site Pain (General disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2) — includes Administration Site Conditions
Catheter Site Inflammation (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) — includes Administration site Conditions
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) — includes Administrations Site Conditions
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a publication (e.g., in a scientific journal) based on the results of this study is envisaged, approval from AstraZeneca will be obtained and a draft manuscript will be submitted to AstraZeneca for scrutiny and comment. The choice of conduit will be mutually agreed on by the Principal Investigator and AstraZeneca.